CLINICAL TRIAL: NCT05885399
Title: A Study on the Efficacy and Safety of Penpulimab in the Treatment of Metastatic Pheochromocytoma/Paraganglioma Patients Who Fail to Other Systemic Treatment
Brief Title: The Efficacy and Safety of Penpulimab in the Treatment of Metastatic PPGL Patients Who Fail to Other Systemic Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06086-06
Record Dates: First submitted 2023-05-22; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Pheochromocytoma, Metastatic; Pheochromocytoma Malignant; Paraganglioma, Malignant
MeSH Terms: conditions — Pheochromocytoma; Neoplasm Metastasis; Paraganglioma, Extra-Adrenal | interventions — penpulimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- penpulimab (Experimental): Penpulimab will be administered intravenously at a dose of 200 mg every 3 weeks. Treatment continued until the patient exhibited radiographic or clinical disease progression or unacceptable adverse events.
  Interventions: Drug: Penpulimab

INTERVENTIONS:
Drug: Penpulimab — Penpulimab will be administered intravenously at a dose of 200 mg every 3 weeks. Treatment continued until the patient exhibited radiographic or clinical disease progression or unacceptable adverse events.

SUMMARY:
Metastatic pheochromocytoma / paraganglioma (MPP) are rare while the prognosis was poor. Penpulimab is specifically an immune check-point inhibitor of PD1 and has been approved for the treatment of several malignancies.This phase II trial studies the efficacy and safety of penpulimab in the treatment of MPP patients who fail to other systemic therapy.

DETAILED DESCRIPTION:
This was a prospective observational study. Patients with histologically or radiologically confirmed MPP and fail to other systemic therapy were enrolled. Penpulimab will be administered intravenously at a dose of 200 mg every 3 weeks. Treatment continued until the patient exhibited radiographic or clinical disease progression or unacceptable adverse events.Plasma normetanephrine and metanephrine (MNs), 24-hour urinary catecholamine excretion (24hCA) were measured at baseline and every 1-3cycle. Contrast-enhanced computed tomography(CT) of chest, abdomen and pelvis were used to assess measurable target lesions at baseline and every 3 cycles. For patients who only had bone metastases or no measurable target lesions, The efficacy was evaluated by 18F-fluorodeoxyglucose (18F-FDG-PET/CT). The primary endpoint was objective response rate (ORR) and the disease control rate (DCR) per Response Evaluation Criteria In Solid Tumors(RECIST) 1.1/PERCIST1.0. Secondary endpoints included biochemical (catecholamine levels) response rate (BRR), progression-free survival (PFS) and safety.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent.
* Age 18-75 years old
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Patients with histologically or radiologically confirmed MPP and fail to other systemic therapy.
* Estimated life expectancy longer than 6 months.
* Confirmed non-pregnancy and lactation. During the entire study period and within 6 months after the last administration, the subjects and their spouses are willing to use efficient contraceptive measures.
* Laboratory requirements:

  * Absolute granulocyte count (AGC) greater than 1.5 x 109/L;
  * Platelet count greater than 80 x 109/L;
  * Hemoglobin greater than 90g/L;
  * Serum bilirubin less than 1.5 x upper limit of normal (ULN);

    --)Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than 2.5 x ULN;
  * Serum creatinine less than 1.5 x ULN or creatinine clearance (CCr)≥60ml/min;
  * Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ lower limit of normal value (50%).

Exclusion Criteria:

* Patients who had been previously treated with anti-PD1, anti-PD-L1, or anti-PD-L2 medications were excluded from this trial.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of trial treatment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has an active infection requiring systemic therapy.
* Didn't meet eligibility for organ function.
* Abnormal coagulation (INR >1.5 or prothrombin time (PT) > ULN 4 seconds or APTT >1.5 ULN), bleeding tendency or being treated with thrombolytic or anticoagulant therapy.
* Uncontrolled congestive heart failure .

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
The objective response rate (ORR) | At the end of Cycle 3(each cycle is 21 days)
  Defined for all patients whose tumor met the criteria of Complete Response (CR)and Partial Response (PR)
The disease control rate (DCR) | At the end of Cycle 3(each cycle is 21 days)
  Defined for all patients whose tumor met the criteria of CR or PR or stable disease(SD)

SECONDARY OUTCOMES:
progression-free survival (PFS) | At least 1 cycle(each cycle is 21 days)
  PFS is defined as the time from the first day of treatment to the first documented disease progression per RECIST 1.1 criteria. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria.
biochemical response | At the end of Cycle 3 (each cycle is 21 days)
  An effective response of 24hCA, MNs or NSE meant that the concentration decreased by more than 40% than the baseline value or decreased to the normal range
Incidence of adverse events | At the end of Cycle 1 (each cycle is 21 days)
  Incidence of adverse events assessed by Common Terminology Criteria for Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Anli Tong, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China